CLINICAL TRIAL: NCT04166357
Title: Early Prediction of Respiratory and Autonomic Complications of GBS Using Neuromuscular Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 5
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Guillain Barre Syndrome
Keywords: Guillain Barre Syndrome, neuromuscular ultrasound
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respiratory and autonomic complications of GBS: Early detection of respiratory failure is among the main challenges raised by the management of GBS. Careful monitoring by an experienced team of nurses and physicians is crucial. The classic signs of respiratory failure occur late, and the early manifestations consist only of tachypnea, tachycardia, air hunger, broken sentences, and a need to pause between sentences; later, use of the accessory respiratory muscles, paradoxical breathing, and orthopnea indicate severe diaphragmatic weakness.
  Autonomic dysfunction occurred in the affected patients, including cardiac arrhythmia, hypertension or hypotension, ileus, and urinary retention.
  Interventions: Diagnostic Test: neuromuscular ultrasound

INTERVENTIONS:
Diagnostic Test: neuromuscular ultrasound — Neuromuscular ultrasound refers to a field in medicine in which ultrasound is used to diagnosis and guide treatment for people with neuromuscular diseases. Neuromuscular ultrasound is often combined with electrodiagnosis, and particularly nerve conduction studies and EMG, to improve the accuracy of diagnosis and add anatomic information to the functional information obtained with electrodiagnosis. It has been demonstrated that neuromuscular ultrasound adds value to the diagnosis of nerve disease in over 80% of cases.

SUMMARY:
Neuromuscular US will be a good and non invasive predictor for respiratory and autonomic dysfunctions in GBS through evaluation of diaphragmatic thickness, phrenic and vagus nerve cross sectional area.

DETAILED DESCRIPTION:
Patients presented in the ER with clinical manifestations and examination suggesting GBS are admitted to neurology department. Confirmation of the diagnosis of GBS is done by fulfilling the clinical diagnostic criteria, CSF examination is done searching for cytoalbuminous dissociation ,serum electrolytes, toxicological screening ,virology to exclude mimics of GBS.

Patients will undergo electrophysiological study (motor NCS of both median ulnar ,tibial ,and peroneal nerves ). Distal motor latency (dmL), nerve conduction velocity (CV) and compound muscle action potential (CMAP)amplitude measurements were undertaken as well as measurements of the mean F-M-latencies of both median ,ulnar and tibial nerves (F-wave latency-dmL). Similarly, sensory nerve conduction study is applied on both median and ulnar nerves ,(dml is assessed. According to the electophysiological study results, patients will be grouped into:

* AIDP: If two or more nerves showed demyelinating features (distal latency prolongation, slow nerve conduction velocity, conduction block, or prolonged F wave latency) on motor nerve conduction study.
* AMAN: Normal sensory conduction studies and unrecordable or reduced compound muscle action potential on motor nerve conduction study. There should not be more than one demyelinating feature in any nerve.
* AMSAN: If both motor and sensory nerve conduction studies revealed features of axonal neuropathy such as reduced or absent CMAP and SNAP, marginal slowing or normal conduction velocity and absence of conduction block.
* Inexcitable: Absent CMAP in all motor nerves (or present in only one nerve with CMAP <10%of lower limit of normal).
* Equivocal: GBS patients not fulfilling the above neurophysiologic criteria.

Then patients will be assessed clinically using the Medical Research Council (MRC) grading for power and Hughes functional grading scale scores.

Muscle groups (right and left) assessed in the measurement of the MRC sums core are:

* Abduction of the arm
* Flexion of the forearm
* Extension of the wrist
* Flexion of the leg
* Extension of the knee
* Dorsal flexion of the foot 0 = No visible contraction

  1. = Visible contraction without movement of the limb
  2. = Movement of the limb but not against gravity
  3. = Movement against gravity over (almost) the full range
  4. = Movement against gravity and resistance
  5. = Normal The MRC-sums core ranges from 0 (paralytic) to 60 (normal strength). (Kleyweg RP et al.,1988)

Guillain-Barré syndrome disability scale 0 A healthy state

1. Minor symptoms and capable of running
2. Able to walk 10 m or more without assistance but unable to run
3. Able to walk 10 m across an open space with help
4. Bedridden or chair bound
5. Requiring assisted ventilation for at least part of the day
6. Dead

Basal and every day arterial blood gases unless new respiratory event occurs. Basal pulmonary function test is done. Clinical assessment for autonomic dysfunction: In addition to reported or clinically evaluated symptoms (sweating problems, orthostatic dysregulation, sexual dysfunction). ECG is done day after day and blood pressure measurements five times daily for at least the first seven days of acute hospitalization.

Ultrasonography is done on diaphragm, phrenic nerve and vagus nerve. As regard diaphragmatic ultrasound:

the index test (ultrasound imaging of the diaphragm) is used. A high-resolution portable ultrasound machine is used, with a 7- to 13-MHz linear array transducer. Patients will be examined in the supine position. The diaphragm was identified as a 3-layered structure lying deep to the intercostals muscles and subcutaneous tissue. 3 images captured at end-expiration and 3 images captured after the patient is asked to inhale as deeply as possible. The transducer is positioned in a sagittal oblique plane, spanning 2 ribs, at approximately the anterior axillary line, overlying one of the most caudal intercostal spaces. Measurements of diaphragm thickness are made using electronic calipers, and the 3 images for each position are then averaged to give a thickness at resting end-expiration (TMIN) and at maximal inspiration (TMAX), from which a diaphragm thickening ratio is derived: TMAX/TMIN. Normal diaphragm thickness is defined as ≥0.14 cm and the normal diaphragm thickening ratio is defined as ≥1.2.

As regard phrenic nerve US:

Under the guidance of a high resolution ultrasound with the patient's head towards the left, the ultrasound probe (frequency, 7-13MHz) was placed on the right side of the neck. The axial scanning of the neck along the surface of the anterior scalene muscle, showed that the phrenic nerve rounded the anterior scalene muscle from the outside to the inside, and coursed through the trench between the common carotid artery and anterior scalene muscle.

As regard vagus us:

All participants were examined with HRUS by a(7-12) MHz transducer. Each VN was visualized in the axial plane at the level of the thyroid gland, and three images were recorded at each side. To assess the VN-CSA its contour within the hyperechoic epineural rim was outlined.. The median of the three VN-CSA measurements was used for statistical analyses.

Patients then undergo plasmapharesis 50 mL/kg, on 5 separate occasions over 1-2 weeks.

Patients after that are evaluated again (4 weeks from the onset of the condition)ie at the end of the acute stage of Guillan Barre syndrome by MRC and Hughes clinical scores and clinical evaluation of autonomic and respiratory dysfunctions will be also assessed . Ultrasound will be done on diaphragm, phrenic nerve and vagus nerve again.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will fulfill the published diagnostic criteria of GBS.
* Age: 18-65
* Both sexes

Exclusion Criteria:

* History of cardiopulmonary dysfunction
* BMI>30 Kg/m2
* Renal or hepatic failure
* Sepsis
* Autonomic or respiratory dysfunction from the start
* Patients with hypo- or hyperkalemic paralysis, porphyria, viral myositis, botulism, diphtheritic neuropathy, and history of potential toxic exposure were excluded.
* Abnormal pulmonary function test from the start.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 Patients that will fulfill the published diagnostic criteria of GBS.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular ultrasound | 24-48 hours
  Sensitivity and specificity of US in predicting respiratory and autonomic complications in Guillain Barre Syndrome

SECONDARY OUTCOMES:
Respiratory and autonomic complications | 1 month
  Incidence of cases developing respiratory and autonomic complications through the course of the disease.
Correlation between clinical scores and reference US values | 48-72 hours
  Correlation between clinical scores and reference US values of diaphragm, phrenic and vagus nerves in prediction of respiratory and autonomic complications of Guillain Barre Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No